CLINICAL TRIAL: NCT01689922
Title: The Effectiveness of Anti-Gravity Treadmill Training in Patients After Lumbar Microdiscectomy and Fusion Surgeries
Brief Title: The Effectiveness of Anti-Gravity Treadmill Training
Status: Terminated | Type: Observational
Why Stopped: slow enrollment
Sponsor: Justin Parker Neurological Institute (Other)
Responsible Party: Sponsor
Other Study IDs: JPNI-2
Record Dates: First submitted 2012-06-12; First posted 2012-09-21 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Lumbar Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- AlterG and Physical therapy: 2) Standard postoperative rehabilitation program with addition of lower body positive pressure (LBPP) treadmill training
  Interventions: Other: AlterG
- Control group: 1) Standard postoperative rehabilitation program
  Interventions: Other: AlterG

INTERVENTIONS:
Other: AlterG — All patients will begin an early postoperative rehabilitation program and standard PT no later than 4 weeks following surgery and continue for at least 6 weeks. The duration of standard PT program could be extended depending on the patient needs. The patients randomized to undergo (LBPP) treadmill training will have an additional 7-week 3 times a week training on the antigravity

SUMMARY:
The primary objective of this study is to compare the effectiveness of standard for our practice postoperative physical therapy (PT) program to a PT program that incorporates lower body positive pressure (LBPP) treadmill training for the patients after lumbar discectomy and fusion surgeries.

DETAILED DESCRIPTION:
A prospective, randomized, parallel group controlled clinical study is proposed. The patients will be divided into the two study groups according to the surgical procedure:

1. patients undergoing one-level microdiscectomy for lumbar herniated disc
2. patients undergoing one-level lumbar fusion for degenerative disc disease without notable spinal stenosis.

Each group will consist of 60 patients (see sample size calculations below) who will be randomized into the two equal groups to undergo:

1. Standard postoperative rehabilitation program
2. Standard postoperative rehabilitation program with addition of lower body positive pressure (LBPP) treadmill training

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 65 years old
* Willing and able to comply with protocol and PT requirements
* Patients with primarily radicular and back pain due to degenerative disc disease requiring one-level discectomy for herniated disc or lumbar fusion between L2 and S1
* Willing and able to sign a study specific informed consent

Exclusion Criteria:

* Require more than one-level surgery
* No previous lumbar surgery
* Any ongoing health condition that would make it difficult to adhere to postoperative PT requirements
* Peri-operative or post-operative complications (infection, pneumonia, nerve injury, dural tear, etc.) that would constraint or delay the ability to participate in postoperative PT
* BMI greater than 40
* Active local or systemic infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing one-level microdiscectomy or fusion surgeries
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2012-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Questionnaire | 24 months
  10 points or 20% improvement on Oswestry Disability Questionnaire

SECONDARY OUTCOMES:
Patient Global Outcome Ratings and Health Quality Improvement | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Alan T Villavicencio, MD, Principal Investigator — Boulder Neurosurgical Associates
Locations (1):
- Boulder Neurosurgical Associates, Boulder, Colorado, United States